CLINICAL TRIAL: NCT05766410
Title: A Randomized, Open-label, Parallel-group Study Comparing the Immune Modulation Effect of Ribociclib, Palbociclib, and Abemaciclib in Early ER+/HER2- Breast Cancer
Brief Title: A Randomized Study Comparing the Immune Modulation Effect of Ribociclib, Palbociclib, and Abemaciclib in ER+/HER2- EBC
Acronym: ORACLE-RIPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202207200MIPB
Record Dates: First submitted 2023-02-03; First posted 2023-03-13 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer; Hormone Receptor-positive Breast Cancer; Hormone Therapy
Keywords: CDK4, 6 inhibitor; Neoadjuvant therapy; Hormone therapy; Hormone Receptor-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; ribociclib; abemaciclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Palbociclib/Letrozole (Experimental): CDK4, 6 inhibitor and endocrine therapy
  Interventions: Drug: Palbociclib; Drug: Letrozole
- Ribociclib/Letrozole (Active Comparator): CDK4, 6 inhibitor and endocrine therapy
  Interventions: Drug: Ribociclib; Drug: Letrozole
- Abemaciclib/Letrozole (Active Comparator): CDK4, 6 inhibitor and endocrine therapy
  Interventions: Drug: Abemaciclib; Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib — CDK4, 6 inhibitor
  Other Names: Ibrance
  Arms: Palbociclib/Letrozole
Drug: Ribociclib — CDK4, 6 inhibitor
  Other Names: Kisqali
  Arms: Ribociclib/Letrozole
Drug: Abemaciclib — CDK4, 6 inhibitor
  Other Names: Venizio
  Arms: Abemaciclib/Letrozole
Drug: Letrozole — Endocrine therapy
  Other Names: Femara

SUMMARY:
The 3 FDA-approved CDK4, 6 inhibitors, palbociclib, ribociclib, and abemciclib, all provided progression-free survival benefits when combined with endocrine therapy in advanced ER+/HER2- breast cancer. But, not all of them provided overall survival benefit in the same setting. One of the proposed mechanisms that influence the overall survival difference is from the different influence of the 3 CDK4, 6 inhibitors on tumor microenvironment and/ or immune system. However, there was no head-to-head comparison of the 3 CDK4, 6 inhibitors in the same study. Neoadjuvant therapy provides a window to obtain tissue samples before treatment, during treatment, and after treatment. We aim to compare the immune modulation effects of palbociclib, ribociclib, and abemaciclib with letrozole in neoadjuvant treatment for ER+/HER2- early breast cancer.

DETAILED DESCRIPTION:
The 3 FDA-approved CDK4, 6 inhibitors, palbociclib, ribociclib, and abemciclib, all provided progression-free survival benefits when combined with endocrine therapy in advanced ER+/HER2- breast cancer. But, not all of them provided overall survival benefit in the same setting. One of the proposed mechanisms that influence the overall survival difference is from the different influence of the 3 CDK4, 6 inhibitors on tumor microenvironment and/ or immune system. However, there was no head-to-head comparison of the 3 CDK4, 6 inhibitors in the same study. Neoadjuvant therapy provides a window to obtain tissue samples before treatment, during treatment, and after treatment. We aim to compare the immune modulation effects of palbociclib, ribociclib, and abemaciclib with letrozole in neoadjuvant treatment for ER+/HER2- early breast cancer. We will collect tumor tissue, blood, and stool samples prospectively before treatment, at 2 weeks after treatment, and after 12 weeks of treatment at the time of surgery. Immune modulation effects will be compared between 3 treatment groups from breast tumor RNAseq analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 20 years old at the time of informed consent.
* Patient has a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer based on the most recently analyzed tissue sample and all tested by local laboratory. with estrogen receptor positive (>10%) on IHC staining and HER2 negative (IHC 0+/1+, or IHC 2+ plus FISH negative)
* Stage II to III
* With adequate organ function
* ECOG 0-1

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless using highly effective methods of contraception during study drug dosing and for 12 months post-dosing
* Patients with active systemic infections or known to have AIDS or to test positive for HIV antibody at Screening
* Any other disease or condition that could interfere with participation in the study according to the study protocol, or with the ability of the patients to cooperate and comply with the study procedures.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The expression of immune-related signature change after different CDK4/6 inhibitor treatments by RNAseq | Through study completion, an average of 3 years
  Characterization of RNAseq from serial tumor biopsy samples

SECONDARY OUTCOMES:
Adverse events | 4 months
  According to CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Department of Oncology, National Taiwan University Hospital, Taipei
  - Department of Oncology,National Taiwan University Hospital, Taipei